CLINICAL TRIAL: NCT06983171
Title: Real-World Clinical Practice Study on the Effectiveness of Semaglutide Over 154 Weeks in Patients With Metabolic Dysfunction-Associated Fatty Liver Disease
Brief Title: Semaglutide Effectiveness in Patients With Metabolic Dysfunction-Associated Fatty Liver Disease in the Real World Practice
Status: Active, not recruiting | Type: Observational
Sponsor: Center of target therapy (Other)
Responsible Party: Sponsor
Other Study IDs: CTT-003
Record Dates: First submitted 2025-04-22; First posted 2025-05-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-05

CONDITIONS: MAFLD
Keywords: CTT-003; Semaglutide in MAFLD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MAFLD patients: * Body mass index (BMI) >30 kg/m².
  * CAP score >238 dB/m (measured by steatometry no more than 3 months before study enrollment).
  * Age 18-70 years at the time of signing informed consent.

SUMMARY:
This real-world clinical trial evaluates the effectiveness of semaglutide (target dose is 2.4 mg/week) over 154 weeks (3 years) prescribed to the patients with metabolic dysfunction-associated fatty liver disease (MAFLD) and liver fibrosis (stages 0-4) as a part of routine clinical practice. MAFLD is a common liver condition linked to obesity, type 2 diabetes (T2DM), and metabolic syndrome, which can progress to severe liver damage (cirrhosis) and heart disease. Currently, there are no approved medications for MAFLD, and treatment relies on lifestyle changes. Semaglutide, a GLP-1 receptor agonist, has shown promise in improving liver health and metabolic markers in earlier studies.

DETAILED DESCRIPTION:
- What is this study about?

This real-world clinical trial evaluates the effectiveness of semaglutide (in target dose of 2.4 mg/week) over 154 weeks (3 years) prescribed to the patients with metabolic dysfunction-associated fatty liver disease (MAFLD) and liver fibrosis (stages 0-4) as a part of routine clinical practice.. MAFLD is a common liver condition linked to obesity, type 2 diabetes (T2DM), and metabolic syndrome, which can progress to severe liver damage (cirrhosis) and heart disease. Currently, there are no approved medications for MAFLD, and treatment relies on lifestyle changes. Semaglutide, a GLP-1 receptor agonist, has shown promise in improving liver health and metabolic markers in earlier studies.

- Why is this study important? MAFLD affects 24% of adults globally, with 20% progressing to advanced stages (MASH/cirrhosis).

MAFLD increases risks of liver failure, cardiovascular disease, and is a leading cause for liver transplants.

- Semaglutide may help by: Reducing liver fat and inflammation. Improving weight, blood sugar, and cholesterol. Slowing liver fibrosis progression.

* Study Details Participants: 70 adults with MAFLD and liver fibrosis (stages 0-4).
* Treatment: Semaglutide (target dose is 2.4 mg/week; however, the dose may be lower in case of poor tolerance or safety concerns).
* Duration: 154 weeks.
* Assessments:

Liver biopsies (to measure inflammation/fibrosis). MRI and elastography (non-invasive liver fat/stiffness tests). Blood tests (liver enzymes, cholesterol, HbA1c). Weight and cardiovascular health monitoring.

- Patient Participation Patients will attend the clinic per the routine clinical practice (it is anticipated that there will be approx. 10 visits over 3 years, with phone check-ins between visits).

Treatment will be conducted in accordance with the local label and routine clinical practice.

* Potential Benefits Access to a promising therapy for MAFLD. Close monitoring of liver and metabolic health. Contribution to advancing MAFLD treatment options.
* Risks and Considerations Semaglutide may cause nausea, diarrhea, or other side effects (typically mild). Liver biopsy carries minimal risks (e.g., pain, bleeding).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before performing any research-related action. Research-related procedures include any procedures conducted within the framework of this study, including activities to assess eligibility criteria for participation in the study.
* Body Mass Index (BMI) > 30 kg/m².
* CAP test result > 238 dB/m based on steatometry performed no later than 3 months before the patient is included in the study.
* Age 18-70 years at the time of signing the informed consent.

Exclusion Criteria:

* Any contraindication to the appointment of semaglutide.
* Documented reasons for chronic liver disease other than non-alcoholic fatty liver disease (NAFLD).
* Positive test result for HBsAg, HIV antibodies, or positive test result for HCV-RNA.
* Presence of ascites, bleeding from esophageal varices, hepatic encephalopathy, spontaneous bacterial peritonitis, or liver transplantation at the time of screening or a history of these conditions.
* ALT activity > 5 times the upper limit of normal (ULN).
* AST activity > 5 times the ULN.
* Alkaline phosphatase activity > 2 times the ULN at screening.
* International Normalized Ratio (INR) of prothrombin time ≥ 1.35 at screening.
* MELD score > 12 points at screening.
* Platelet count less than 150,000 per microliter of blood, unless it reflects the patient's usual platelet level, and the patient does not have a diagnosis of portal hypertension in the investigator's opinion.
* Treatment with GLP-1 receptor agonists within 90 days prior to the screening visit.
* Treatment with hypolipidemic drugs or weight loss medications, whose dosage has not been stable, in the investigator's opinion, for 90 days prior to the screening visit.
* Previous or planned (during the study period) treatment of obesity with surgical intervention or the installation of a special device for weight loss. However, the following procedures are allowed:

  1. Liposuction and/or abdominoplasty, if performed more than 1 year before screening.
  2. Laparoscopic gastric banding, if the band was removed more than 1 year before baseline liver biopsy and screening.
  3. Intragastric balloon placement, if the balloon was removed more than 1 year before baseline liver biopsy and screening.
  4. Duodenojejunal sleeve bypass, if the sleeve was removed more than 1 year before baseline liver biopsy and screening.
* Presence of malignant neoplasms currently or in history within the last 5 years prior to screening. Exceptions include only basal cell or squamous cell skin cancer and any carcinoma in situ.
* History of acute pancreatitis within 180 days prior to inclusion in the study.
* Presence of chronic pancreatitis currently or in history.
* Any of the following: myocardial infarction, stroke, heart failure of NYHA class IV, hospitalization for unstable angina, or transient ischemic attack within the last 90 days before the screening day.
* Any health disorder that, in the investigator's opinion, could jeopardize patient safety or affect compliance with the protocol requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adults aged 18-70 years with obesity (BMI >30 kg/m²) and hepatic steatosis (CAP >238 dB/m) confirmed within 3 months. Eligible participants must have metabolic dysfunction-associated fatty liver disease (MAFLD) without other chronic liver conditions (e.g., viral hepatitis, cirrhosis complications like ascites, or MELD score >12).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2028-09-12 (Estimated); Study Completion 2028-09-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of semaglutide therapy on liver morphological changes based on liver histology using the NAFLD Activity Score (NAS). | 154 weeks
  To compare change in the degree of steatosis, severity of inflammation, ballooning degeneration, stage of fibrosis NAFLD Activity Score (NAS = 0-8 points) at the end of treatment relative to baseline values
Evaluate the impact of semaglutide therapy on the degree of steatosis change based on Controlled Attenuation Parameter (CAP score) | 154 weeks
  Evaluate the degree of liver steatosis change based on the CAP test in dB/m at the end of treatment relative to the baseline value
Evaluate the impact of semaglutide therapy on the degree and distribution of fat infiltration in the liver based on MR spectroscopy data | 154 weeks
  Change in the quantitative data on the content and distribution of fat in the liver at the end of treatment relative to the baseline value
Evaluate the impact of semaglutide therapy on changes in liver elasticity based on elastography data | 154 weeks
  Change in liver fibrosis stage based on elastography data (kPa) at the end of treatment relative to the baseline value

SECONDARY OUTCOMES:
Evaluate the impact of semaglutide therapy on patients' body weight | 154 weeks
  Change in percentage of patients' body weight at the end of treatment relative to the baseline value
Evaluate the impact of semaglutide therapy on changes in aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels | 154 weeks
  Change in ALT and AST activity (measured in U/L) at the end of treatment relative to the baseline value
Evaluate the impact of semaglutide therapy on changes in Total Cholesterol, Low-Density Lipoprotein (LDL) Cholesterol, High-Density Lipoprotein (HDL) Cholesterol and Triglycerides levels | 154 weeks
  Сhanges in Total Cholesterol, Low-Density Lipoprotein (LDL) Cholesterol, High-Density Lipoprotein (HDL) Cholesterol and Triglycerides levels (in mmol/L) at the end of treatment in comparisson with the baseline values
Evaluate the impact of semaglutide therapy on changes in High-sensitivity C-reactive Protein (hs-CRP) level | 154 weeks
  Сhanges in High-sensitivity C-reactive Protein (hs-CRP) level (in mg/L) at the end of treatment in comparisson with the baseline values
Evaluate the time to the first cardiovascular event during semaglutide therapy | 154 weeks
  Time to first serious cardiac and hepatic event in days from the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Bogomolov, Prof., PhD, MD, Principal Investigator — Center of target therapy
Locations (1):
- Center of Target Therapy LLC., Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided